CLINICAL TRIAL: NCT06385912
Title: Systematic Lymphadenectomy During Interval Debulking Surgery in Advanced Epithelial Ovarian Cancer: a Multicenter Real-world Study
Brief Title: Systematic Lymphadenectomy During Interval Debulking Surgery in Advanced Epithelial Ovarian Cancer
Status: Completed | Type: Observational
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Qinglei Gao, Professor, Tongji Hospital
Other Study IDs: 2024-TJ-SLIDS
Record Dates: First submitted 2024-04-20; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Ovarian Cancer; Postoperative Complications; Neoadjuvant Therapy; Lymph Node Excision
Keywords: Advanced epithelial ovarian cancer; Lymphadenectomy; Neoadjuvant chemotherapy; Interval debulking surgery; Prognosis; Postoperative complication
MeSH Terms: conditions — Ovarian Neoplasms; Postoperative Complications | interventions — Lymph Node Excision

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lymphadenectomy group: Patients received lymphadenectomy during IDS
  Interventions: Procedure: lymphadenectomy
- no lymphadenectomy group: Patients did not receive lymphadenectomy during IDS

INTERVENTIONS:
Procedure: lymphadenectomy — Systematic pelvic and para-aortic lymphadenectomy during IDS in lymphadenectomy group
  Groups: lymphadenectomy group

SUMMARY:
The study aims to investigate the prognostic and postoperative complication relevance of lymphadenectomy in advanced epithelial ovarian cancer patients who received neoadjuvant chemotherapy (NACT) followed by interval debulking surgery (IDS). The main question it aims to answer is:

Does systematic lymphadenectomy during interval debulking surgery have a significant impact on survival in patients with advanced epithelial ovarian cancer who have received neoadjuvant chemotherapy?

The progression-free survival (PFS), overall survival (OS), and postoperative complication were compared between the lymphadenectomy and no lymphadenectomy groups to answer the question.

DETAILED DESCRIPTION:
The study aims to investigate the prognostic and postoperative complication relevance of lymphadenectomy in advanced epithelial ovarian cancer patients who received neoadjuvant chemotherapy (NACT) followed by interval debulking surgery (IDS). The study included patients with histologically confirmed advanced epithelial ovarian cancer who received IDS at seven tertiary hospitals in China from 2006 to 2021. The progression-free survival (PFS), overall survival (OS), and postoperative complication were compared between the lymphadenectomy and no lymphadenectomy groups. Propensity score matching (PSM) and overlapping weight (OW) analyses were performed to minimize selection bias.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients with advanced epithelial ovarian cancer (stage IIB-IV, according to the International Federation of Gynecology and Obstetrics (FIGO) 2014);
2. Patients who underwent NACT followed by IDS.

Exclusion Criteria:

1. Patients with early-stage ovarian cancer (FIGO stage I-IIA);
2. Patients only receiving primary debulking surgery (PDS) as initial treatment without NACT;
3. Histological subtypes other than advanced epithelial ovarian cancer;
4. Patients with unclear sites of lymphadenectomy and non-compliant systematic lymphadenectomy that not include pelvic and/or para-aortic lymph nodes.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 1090 patients diagnosed with FIGO stage IIB-IV epithelial ovarian cancer and who underwent IDS following NACT were selected for eligibility from July 2006 to February 2021 based on the NUWA Platform from 7 centers. Twenty-two patients who had unclear and non-compliant systematic lymphadenectomy were excluded and 1068 patients were enrolled in this study. Out of these patients, 528 (49.4%) had an IDS with lymphadenectomy, while 540 (50.6%) had an IDS without lymphadenectomy.
Sampling Method: Probability Sample
Enrollment: 1090 (Actual)
Dates: Start 2006-07-01 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From the initial diagnosis to the occurrence of recurrence, progression, death, or the latest follow-up, whichever came first, until February 10, 2021, an average of 3 years
  The progression-free survival (PFS) was defined as the duration from the initial diagnosis to the occurrence of recurrence, progression, death, or the latest follow-up, whichever came first.
Overall survival (OS) | From the initial diagnosis to the occurrence of recurrence, progression, death, or the latest follow-up, whichever came first, until February 10, 2021, an average of 5 years
  Overall survival (OS) was described as the duration from the date of diagnosis to the date of death from any cause or the last follow-up date.

CONTACTS AND LOCATIONS:
Overall Officials: Qinglei Gao, MD, PhD, Study Chair — Tongji Hospital
Locations (1):
- Tongji Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided